CLINICAL TRIAL: NCT06276751
Title: The Diagnostic Value of End-Tidal CO2 in Patients Diagnosed With Pneumothorax in the Emergency Department and Its Role in Predicting Patient Outcomes
Brief Title: The Diagnostic Value of End-Tidal CO2 in Patients Diagnosed With Pneumothorax
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Safa Dönmez, M.D., Ankara City Hospital Bilkent
Other Study IDs: E1-23-3870 ptx endtidalco2
Record Dates: First submitted 2024-02-15; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: End-tidal CO2 monitor — Throughout the study, measurements were taken at 2 and 4 hours after tube thoracostomy was applied to every patient undergoing the procedure.
  Other Names: Measurement of end-tidal CO2 after tube thoracostomy application.

SUMMARY:
Pneumothorax (PTX) is defined as the accumulation of air in the pleural space. PTX can cause a disruption in the perfusion of lung tissue in the affected area and increase intrathoracic pressure, potentially leading to obstruction of venous return and, consequently, posing a life-threatening condition. Therefore, PTX requiring urgent intervention is a significant concern in emergency departments.

End-tidal carbon dioxide (ETCO2) provides insight into carbon dioxide levels resulting from lung perfusion and serves as a respiratory parameter informing the prognosis of various critical illnesses. One of the most important factors determining lung perfusion is the effective lung area. Among the crucial issues for emergency departments are PTX cases, which typically regress following urgent intervention, leading to the establishment of an effective lung area. Hypotheses have been proposed in the literature suggesting that ETCO2 may be affected in PTX cases due to the relationship between effective lung area and ETCO2.

In this study, investigetors aimed to investigate changes in ETCO2 levels following tube thoracostomy applied to PTX cases.

DETAILED DESCRIPTION:
In the study, a GE brand patient monitor (GE Medical Systems Information Technologies, Germany) was used for vital parameters, and a Medtronic brand Capnostream 35 respiratory monitor device (Oridion Medical 1987 Ltd., Israel) was used for ETCO2 measurement. Patients' ETCO2 measurements were performed using a device that measures ETCO2 levels in breaths delivered through the mouth and nose (sidestream measurement). ETCO2 values were measured before tube thoracostomy placement and at 2 and 4 hours after placement. The diagnosis of pneumothorax was confirmed by chest X-ray. Tube thoracostomy was performed by chest surgeons or emergency physicians. Indications for tube thoracostomy were determined by chest surgery doctors.

Patients' age, gender, height, weight, vital signs, smoking history, pneumothorax causes, lateral and apex collapse amount (in mm), procedures performed, ETCO2 values before and after tube insertion at 2 and 4 hours, hemogram, biochemistry, and blood gas values were recorded on case report forms. Additionally, patients' lengths of stay were recorded using archive numbers through the hospital automation system.

On chest X-ray, a distance greater than 2 cm between the parietal and visceral pleura at the hilum level according to British guidelines or a distance greater than 3 cm from the apex according to American guidelines was defined as a large pneumothorax. Additionally, the percentage of PTX volume for patients was calculated using the Collins method. The PTX percentage was calculated using the formula "%Collins = '4.2 + 4.7(a + b + c)'", where 'a' is the maximum apical interpleural distance, 'b' is the interpleural distance at the midpoint of the upper half of the lung, and 'c' is the interpleural distance at the midpoint of the lower half of the lung.

Neutrophil Lymphocyte Ratio (NLR) and Platelet Lymphocyte Ratio (PLR) calculations were performed.

The initial ETCO2 (ETCO2-0) was defined as the ETCO2 measured at the emergency department visit. PaCO2 was defined as the partial pressure of carbon dioxide measured with the first blood gas analysis taken at the emergency department visit. After lung expansion, ETCO2 was defined as the average value of ETCO2 measured 2 to 4 hours after tube thoracotomy (ETCO2-1/ETCO2-2, respectively). The increase in ETCO2 after expansion was defined as the increase in ETCO2 after closed tube thoracotomy (ETCO2 increase after drainage = ETCO2 after tube thoracotomy - initial ETCO2). The change from ETCO2-0 to ETCO2-1 was determined as deltaETCO2-1 (ΔETCO2-1), and the change from ETCO2-0 to ETCO2-2 was determined as ΔETCO2-2.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Individuals without comorbidities
* Those diagnosed with spontaneous or traumatic pneumothorax
* Patients who underwent tube thoracostomy
* Individuals without other organ damage or injury

Exclusion Criteria:

* Patients under 18 years of age or over 65 years of age
* Patients who refuse to participate in the study
* Pregnant women
* Individuals diagnosed with acute/chronic lung disease
* Those with a history of advanced heart failure
* Individuals with advanced systemic disease
* Patients with a history of malignancy (cancer)
* Individuals with chronic liver disease
* Those using sedative and analgesic neuro-psychiatric drugs
* Patients with a history of psychological or neurological disorders
* Individuals with acute organ damage or failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients aged 18 and over, without any comorbidities, diagnosed with spontaneous or traumatic pneumothorax, who underwent tube thoracostomy, and had no other organ damage or injury.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
ETCO2-0 | Five minutes have passed since the emergency room application.
  It was defined as the end-tidal CO2 (ETCO2) measured at the emergency department visit.
ΔETCO2-1 | Two hours after the emergency room application.
  The change in ETCO2-1 compared to ETCO2-0.
ΔETCO2-2 | Four hours after the emergency room application.
  The change in ETCO2-2 compared to ETCO2-0.
ETCO2-1 | Two hours after the emergency room application.
  End-tidal CO2 measured 2 hours after emergency department admission.
ETCO2-2 | Four hours after the emergency room application.
  End-tidal CO2 measured 2 hours after emergency department admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not currently planned.

REFERENCES:
- [Background] Lee GM, Kim YW, Lee S, Do HH, Seo JS, Lee JH. End-Tidal Carbon Dioxide Monitoring for Spontaneous Pneumothorax. Emerg Med Int. 2021 Jun 14;2021:9976543. doi: 10.1155/2021/9976543. eCollection 2021. PMID 34234966